CLINICAL TRIAL: NCT04761042
Title: A Randomized Controlled Pilot Study Assessing Feasibility and Impact of a Wilderness Program on Mental and Physical Health of Adolescent and Young Adult Cancer Survivors
Brief Title: Wilderness Program for Adolescent and Young Adult Cancer Survivors
Acronym: WAYA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid Sweden University (Other)
Collaborators: UiT The Arctic University of Norway (Other); University of California, San Francisco (Other); See You At The Summit (Unknown); Sörlandet Hospital, Norway (Unknown); The Swedish Winter Sports Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Dnr 2019-67
Record Dates: First submitted 2021-01-21; First posted 2021-02-18 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: wilderness therapy; adventure therapy; recreational therapy; outdoor therapy; nature; adolescent; young adult; childhood cancer survivors; health promotion; positive health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A Randomized control design where participants are randomized to one of the two groups, stratification is made for gender and age (older/younger).
Who Masked: Outcomes Assessor
Masking Description: After being screened for recruitment by the primary investigator, participant are randomized into the two group. Randomization is made by a second team member that up till then had no contact with participants or knows their names (based on screening numbers).
  After being notified of groups assignment the primary investigator again contacts participants to enter the into the study and give information on group assignment.
  Outcome data will be entered confidential, and the outcomes assessor will be blinded regarding group assignment and identification of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wilderness program (Experimental): A one-week (8 days) wilderness program, 3-month online support, and a follow-up visit for four days.
  Interventions: Other: WAYA-Wilderness
- Holiday program (Attention control) (Other): A one-week (8 days) holiday program, 3-month online contact, and a follow-up visit for four days.
  Interventions: Other: WAYA-Holiday

INTERVENTIONS:
Other: WAYA-Wilderness — The wilderness intervention includes challenging tasks in order to help participants' overcome and master new physical and psychological challenges in an unknown environment, with the idea to support self-efficacy, self-esteem, and ability to recover from adversity. The program is designed to encourage participants to connect with nature as to experience gratitude for the richness of the natural world, a sense of calmness and trust upon spending time in nature, and to be more physically active in nature.
  Elements previously described Participants will continue in a three-month program at home (on-line supported) after the initial 8-days in order to empower participants to incorporate elements of the onsite wilderness program into their daily life. An individualized a plan for activities will be developed together with the participant.
  After three months, there will be a re-visit with follow up on outcome measures and reconnection.
  Arms: Wilderness program
Other: WAYA-Holiday — An attention control group (information in "Detailed description")
  Arms: Holiday program (Attention control)

SUMMARY:
Young cancer survivors are at higher risk of cancer reoccurrence, frailty, suicidal ideation, sedentary behaviour, reduced quality of life, and reduced overall life expectancy, compared to their siblings or healthy young persons. Development of new interventions after cancer treatment is urgently needed in order to reduce and diminish these unwanted risks in young cancer survivors. Previous studies have reported that wilderness therapy may reduce anxiety/depression, improve body image and self-efficacy, and increase physical activity in young adult cancer survivors.

High quality randomized controlled studies are lacking and thereby urgently needed to investigate the impact of wilderness programs on mental and physical health of adolescent and young adult cancer survivors. The primary aim of this study is to conduct a pilot randomized controlled trial (RCT) on a wilderness program versus an attention-control activity in adolescent and young adult cancer survivors. We will examine the feasibility of performing a RCT and examine health outcomes, in preparation for a larger RCT with adolescent and young adult cancer survivors.

A total of 40 adolescent and young adult cancer survivors (aged 16-39) will be randomized to a wilderness intervention or an attention-control group. The wilderness intervention is a one-week outdoor program where participants have individualized and group activities such as climbing, hiking, kayaking, bush crafting and mindfulness. After this week, participants continue a 3-month program to incorporate elements of the intervention into their daily life. The control group will join a relaxing one-week holiday at a Wellness Center and will be followed for 3 months to control for attention. Study outcomes will be recruitment speed, willingness to be randomized, study adherence, self-reported mental health using validated scales, and tests of physical activity and health (six-minute walk test, submaximal oxygen uptake, blood pressure, sedentary behaviour and physical activity). Outcomes are measured at the start of the study, 1 week and 3 months after intervention. One year follow up of self-reported outcomes will be online. Findings of the study will provide important insights into the feasibility of a large study as well as on ways by which wilderness therapy can promote health in young cancer survivors.

DETAILED DESCRIPTION:
Aim of the study The objective of the present study is to conduct a pilot randomized controlled trial (RCT) on a wilderness program versus an attention-control activity in adolescent and young adult cancer survivors. We will examine the feasibility of performing a RCT, in preparation for a larger RCT with adolescent and young adult cancer survivors, as well as to investigate individuals' experience and safety of the wilderness program. To the best of our knowledge, we are preparing the first RCT that will be undertaken to investigate the impact of a wilderness program in adolescent and young adult cancer survivors.

It is hypothesized that the wilderness program is a highly appreciated and safe health promotion intervention that may substantially benefit adolescent and young adult cancer survivors, and that results of the proposed pilot study warrant further research with adequate power to test for effectiveness in a larger RCT.

RCT - Intake (Contact 1)

Young cancer survivors who are interested in participating will contact the researchers of this study at Mid Sweden University via email or phone. The researchers will provide information about the study, both verbally and written in an information letter to be sent by post or email. The following tasks will be carried out at the intake interview:

* Screening of inclusion and exclusion criteria,
* Explanation/information about the study and informed consent procedures,
* Explanation/information about the interventions and the randomisation procedure,
* Check participants' willingness to be randomized, ask if they have a strong preference for either intervention, and ask about their expectations of the interventions,
* Sending the information letter and informed consent forms, including a postage-paid return envelope.

Randomisation (Contact 2)

Written informed consent from the participants will be obtained prior to randomisation. One of the researchers of this study will also sign the informed consent form. After the signed informed consent form has been received, young cancer survivors will be randomised for participation in the study. All data of each randomized participant in the study will be documented in a Case Report Form (CRF) that will be developed for this study. Participants will be contacted by telephone and the following tasks will be carried out:

* Inform participants about the outcome of the randomisation procedure,
* Collect demographic data (DD), medical history (MH), medication use (MU), concomitant medication/therapies, dietary and lifestyle measures,
* Instructions for using the step counter, one week before the start of intervention: All participants that are randomized in the study will be send a step counter, to be used in the week before the intervention,
* Sending the step counter and instructions for use to participants,
* Instruction for measurements and timelines during the study.

Intervention (Visit 1) All participants will travel for the intervention (8 days in total) to Sundsvall, Sweden. At Day 1 of the intervention (Baseline, T=0), participants will perform physical performance/fitness tests at Mid Sweden University under supervision of a test leader from the Sweden Winter Sports Research Centre (Östersund, Sweden). After the tests, participants in the intervention group will be transported to the wilderness site at Höga Kusten, Västernorrland, Sweden. Participants will be provided with outdoor clothes, backpack, tent, sleeping pads and sleeping bag. All other necessary outdoor equipment will be made available through the facilitators. Participants in the control group will be transported to a Wellness Center in Västernorrland. Before leaving for home, a plan for activities in the three-month home program will be discussed with participants in the wilderness program group.

Three-months at home (Contact 3 and 4)

Participants in both groups will be followed during a 3-month period after the one-week intervention. During this period, participants will be contacted by a facilitator via telephone or other media after one month (Contact 3) and two months (Contact 4). The following tasks will be carried out:

* Documentation of concomitant medication/therapy use, dietary and lifestyle measures,
* Documentation of adverse events that may have occurred,
* Filling in the IPAQ,
* Results of the step counter during the week before Contact 3 and 4,
* Adherence and transference of participants to the agreed and planned activities at home (wilderness program group only).

Intervention (Visit 2; Re-visit) After three months, participants will return to Mid Sweden University for follow up measures (T=2), as well as for two additional nights outdoor at Höga Kusten to re-connect (intervention group) or two holiday nights at the Wellness canter (Control group).

One year follow-up One year after start of the intervention (T=3), participants in both groups will be contacted to fill in online self-reported questionnaires. Concomitant medications/therapies, dietary and lifestyle measures will be documented as well as a recent one-week measurement of step counts.

Sample size No sample size calculation is needed for a pilot RCT.

Randomization Participants will be randomized according to a randomization list as generated by the Random Allocation Software Program using a random block size of 2 in order to guarantee a balanced allocation. The two interventions (wilderness therapy versus attention-control are assigned to intervention A and intervention B and upon intake participants will receive a screening number ranging from 01 to 100. Participants who drop out of the study before being randomized will keep their screening number without receiving an intervention. On enrolment in the study, participants that are randomized receive an intervention number (01-110). The study numbers are sequentially allocated to the participants in the order of inclusion in the randomized intervention period. Each participant will receive only that intervention which is labeled with the study number allocated to him/her. Participants will be stratified according to age group (16-22 and 23-30 and 31-39) and gender (male/female) in order to achieve equal distribution among the two groups. Per stratification, separate randomization lists will be generated.

Statistics Regular descriptive statistics will be calculated with regard to demographical and categorical data and mean scores and standard deviations of the numerical variables will be calculated using SPSS (version 25.0). As a first step, preliminary mean differences between, and within groups (over time changes) will be calculated using students t-test, related samples t-test, and R-ANOVA analysis. As a second step, the Aickin separation test will be applied to the domains of the MMQL and other outcome measures to determine whether there are indications of differences, even if obtained p-values are non-significant. If indications of differences are identified with the Aickin separation test it provides information whether a further larger RCT is warranted. The Aickin separation test is used for early phase trials to determine whether the data are 1) in the hypothesized direction, 2) counter to the hypothesized direction or 3) equivocal. Results in the hypothesized direction warrant further research with adequate power to test for effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Participants of:

* any sex,
* aged 16-39,
* diagnosed with any type of cancer during their course of living
* can be reached by telephone,
* have good understanding of the Swedish language.
* ability to walk 2 km without pausing (walking aids permitted).

Participants with various medical conditions, including mobility impairments, amputees, vision impairments and special treatment or diet needs will be included. No prior experience with any outdoor activity is required.

Exclusion Criteria:

* active cancer treatment for which participation in the study can involve unwanted risks (as evaluated by their treating physician/oncologist),
* other medical conditions that prevent safe travel to, or participation in the program

Ages: 16 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Gender will be expressed in terms of self-representation
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Participant Preferences | At prestudy screening - prior to inclusion
  Participant Preferences (P-Pref) regarding intervention arms (no pref, slight pref, strong preference)
Feasibility - Participant expectations | At prestudy screening - prior to inclusion
  A textual description of what participants would expect to experience from participation in either intervention group.
Feasibility - Participant willingness to be randomized | At prestudy screening - prior to inclusion
  Willingness of participants to be randomized (Yes/No)
Feasibility - Time to recruitment | Until predetermined number of participants are reached or max up till 18 months
  A planned n of 40 is planned and documentation of time to reach the goal will be made until predetermined number of participants are reached or max up till 18 months
Feasibility - Participant Adherence to Protocol | through study completion, an average of 1 1/2 year
  Adherence of the participants to the study protocol. A textual description of participant adherence based on observation and interviews documented in the participants study protocol
Feasibility - Logistics and Burden | Through study completion, an average of 1 1/2 year
  Logistics and Burden (for participants) to perform physical performance/fitness tests. A textual description of participant Log-BurdenPhysbased on observation and interviews documented in the participants study protocol
Feasibility - Logistics and willingness to complete all planned study-related questionnaires | Through study completion, an average of 1 1/2 year
  Logistics and willingness to complete all planned study-related questionnaires. A textual description of participant Log-WillQuest based on observation and interviews documented in the participants study protocol
Feasibility - Adherence to three month at home program | up to three months
  The adherence of the participants to the three months at home program and transference of activities in this period. A textual description of participant adherence based on observation and interviews documented in the participants study protocol
Feasibility - Occurrence of adverse events | up to three months
  Occurrence of adverse events during program execution. A textual description of occurence of AdvEvents based on observation and interviews documented in the participants study protocol.
  Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) and analysed using preferred terms and allocation to system organ class. Safety of the interventions will be measured by analyzing number and type of adverse events reported.

SECONDARY OUTCOMES:
Minneapolis Manchester Quality of Life - MMQL | Baseline, 2 weeks post intervention, 3-month, and 12 month follow up
  Minneapolis Manchester Quality of Life instrument - MMQL, at baseline prior to intervention, prior to 3 month follow up, and after one year.
  The MMQL-Adolescent form is a quality of life questionnaire specifically designed for young cancer survivors (age 13-20 years old) and consists of seven quality of life domains; physical, cognitive, psychological and social functioning, body image, intimate relations, and outlook on life. Scoring on the MMQL ranges from 1 to 5; 5 indicates maximal HRQL. An overall quality-of-life (QOL) score is also computed. Includes 45 items, total sum ranging between 45 and 225 The instruments has good psychometric characteristics and is translated and validated in the Swedish context.
International Physical Activity Questionnaire | Baseline, 2 weeks post intervention, 3-month, and 12 month follow up
  International Physical Activity Questionnaire (IPAQ), at baseline prior to intervention, prior to 3 month follow up, and after one year.
  Subjective reporting of time spent on performing different levels of physical activity, reported in days, hours, and minutes.
  An instrument evaluated as having good psychometric properties, and also translated into Swedish language:
Generalized Self-Efficacy Scale | Baseline, 2 weeks post intervention, 3-month, and 12 month follow up
  Generalized Self-Efficacy Scale (GSE), data collected at baseline prior to intervention, prior to 3 month follow up, and after one year.
  The GSE scale consists of 10 items rated on a four-point (1-4) Likert scale (''not at all true'' to ''exactly true''). Means are calculated as the sum of all answers divided by ten (the total number of items).
  An instrument evaluated as having good/acceptable psychometric properties, and also translated into Swedish language:
Rosenberg Self-Esteem Scale RSES | Baseline, 2 weeks post intervention, 3-month, and 12 month follow up
  Rosenberg Self-Esteem Scale (RSES) at baseline prior to intervention, prior to 3 month follow up, and after one year The scale has four-graded (1-4) Likert-type responses where a rating of one represents the worst and four the best self-esteem. Minimal score10 maximum 40.
  An instrument evaluated as having good psychometric properties, and also translated into Swedish language.
Nature Relatedness Scale | Baseline, 2 weeks post intervention, 3-month, and 12 month follow up
  Nature Relatedness Scale (NRS), at baseline prior to intervention, prior to 3 month follow up, and after one year The scale has 21 items that have five-graded (1-5) Likert-type responses where a rating of one represents the least agreement with item statement and five full agreement. An overall NRS score is calculated where means are calculated as the sum of all answers divided by 21 (the total number of items). The scale also has three subscale that can be extracted and calculated in the same way as the total sum.
  An instrument evaluated as having good psychometric properties in English. Previously not used in Swedish language but now translated and re-translated by the research group and the scale is presently undergoing psychometric testing.
Physical performance - Six Minute Walking Test | Baseline, 3-month
  Six Minute Walking Test - Will be collected during the first day of the 8 day program, and the first day of three month follow up.
  A frequently used test where participant walks on a standardized path, trail, track for six minutes, and the outcome is expressed in number of meters walked.
Physical performance -Oxygen uptake | Baseline, 3-month
  Oxygen uptake - The Ekholm-Bak submaximal test for oxygen (VO2max) uptake will be collected during the first day of the 8 day program, and the first day of three month follow up.
  Outcome- VO2max comprises and is expressed as: L/min, ml/kg/min, but is calculated by combining measures of Maximal heartrate (HRmax) - beats/min, and perceived exertion (Borg Scale 6-20, where a 6 represents a very light exertion and 20 an extremely (too hard) exertion.
  The Ekholm-Bak test is submaximal cycle ergometer aerobic fitness test evaluated as being valid, reliable and safe to use in vulnerable populations.
Heart Rate | Baseline, 3-month
  Heart rate - Resting heart rate (Beat/min) will be recorded during the first day of the 8 day program, and the first day of three month follow up
Blood Pressure | Baseline, 3-month
  BP - Resting systolic and diastolic blood pressure (mmHg) will be recorded during the first day of the 8 day program, and the first day of three month follow up
Physical performance - Level of Physical activity | Baseline, 2 weeks post intervention, 3-month, and 12 month follow up
  Steps - mean steps per day during one week. at baseline prior to intervention, prior to 3 month follow up, and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jong, PhD, Principal Investigator — Dep of Health Sciences/Public Health, Mid Sweden University, Sundsvall, Sweden
Locations (1):
- Mid Sweden University, department of Health Sciences, Sundsvall, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Raw confidential data can be shared upon request after publication in scientific journal
Supporting Information: Study Protocol, ICF
Time Frame: can be shared upon request after publication in scientific journal: Earliest Spring 2024
Access Criteria: By Swedish Law, research data must be provided if authorized researchers request it. By definition that corresponds to someone who has research training and an academic doctoral degree.

REFERENCES:
- [Derived] Jong MC, Dahlqvist H, Lown EA, Schats W, Beckman L, Jong M. A randomized controlled pilot study assessing feasibility and safety of a wilderness program for childhood, adolescent, and young adult cancer survivors: the WAYA study. BMC Public Health. 2023 Aug 8;23(1):1504. doi: 10.1186/s12889-023-16408-x. PMID 37553637
- [Derived] Jong MC, Mulder E, Kristoffersen AE, Stub T, Dahlqvist H, Viitasara E, Lown EA, Schats W, Jong M. Protocol of a mixed-method randomised controlled pilot study evaluating a wilderness programme for adolescent and young adult cancer survivors: the WAYA study. BMJ Open. 2022 May 9;12(5):e061502. doi: 10.1136/bmjopen-2022-061502. PMID 35534081